CLINICAL TRIAL: NCT05013294
Title: Using mHealth to Optimize Glycemic Control in Adults With Type 2 Diabetes in Nakuru County: A Proof-of-Concept Randomized Controlled Trial
Brief Title: Using mHealth (Mobile Health) to Optimize Glycemic Control in Adults With Type 2 Diabetes: Proof of Concept Study
Acronym: mHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology (Other)
Responsible Party: Principal Investigator, Moses Mokaya, PhD Researcher, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P959-2021
Record Dates: First submitted 2021-07-20; First posted 2021-08-19 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Diabetes
Keywords: Type 2 diabetes; mHealth (mobile health); Behavior Change Wheel
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Methods; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive a total of 43 text messages. Text messages were developed using the Behavior Chang Wheel (BCW) through a systematic process linked to specific behavior change techniques. The text messages will provide practical information or guidance to influence selection and eating healthy diet for type 2 diabetes care. The text messages were either loss- or gain-framed to increase influence on behavioral decisions. Additionally, the participants will receive a text message to rate their ability on selection of food and eating of healthy diet based on the messages received in the month. The combination of the one-way and two-way messages in this group are designed to increase engagement of the participants.
  Interventions: Other: Intervention
- Control Arm (Placebo Comparator): The control group will continue receiving standard care in the hospitals. The control group shall also receive a reminder text messages one day prior the routine clinic appointment. The clinic appointment dates shall be derived from the hospital where the participant receives routine diabetes care.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Text messages through a basic phone or smart phone
  Other Names: mHealth

SUMMARY:
The objective of this study is to evaluate the efficacy of a diet-related mHealth (mobile health) intervention on glycated hemoglobin among adults with type 2 diabetes. The study hypothesizes that using mHealth influences food literacy and dietary behavior and may result in a reduction of glycated haemoglobin (HbA1c) by at least 0. 3% in 12 weeks in adults with type 2 diabetes. This study will be conducted in Nakuru County, a cosmopolitan county located in Northwestern Kenya. Participants will be eligible to be included in the study if they will meet the following criteria: (i) adults over the age of 18 years; (ii) diagnosed with type 2 diabetes in the previous 1 year and obtaining care at a participating level 4 hospital; (iii) able to read and write English or Swahili Language; (iv) currently own and able to read and send mobile text messages using any phone. Participants will be excluded if they are on dialysis or pregnant. The primary outcome measure will be HbA1c, which shall be measured at baseline and at the end of the intervention. Secondary outcome measures will include fasting plasma Glucose (FPG), total cholesterol (TC), triglycerides (TG) and high-density lipoprotein-cholesterol (HDL-C). Other secondary outcome measures will include anthropometric measurements (weight, height, waist and hip circumferences) and behaviour change (changes in dietary intake of legumes, fruits and vegetables). Additionally, mHealth satisfaction shall be assessed at 12 weeks and 24 weeks post-intervention to assess the sustainability of the intervention.

DETAILED DESCRIPTION:
A sample size of 60 a-priori (n=30 intervention, n=30 control arm) was determined to assess feasibility of text messaging in optimizing glycemic control. It is anticipated that this proof-of-concept study will obtain parameters that will be used in determining a robust power calculation for a fully powered efficacy trial. Purposive sampling will be used to select two hospitals, one in a rural setting and another in an urban setting in Nakuru County, Kenya. Multistage random sampling using computer-generated list of random numbers will then be applied to randomly assign 15 participants to either the intervention arm or control arm. The hospitals' diabetes registers will be used to select patients on regular diabetes care from the hospital patient records.

The intervention group will receive a total of 43 text messages developed using the Behavior Change Wheel (BCW) approach. The text messages that are linked to specific behavior change techniques will provide practical information or guidance to influence selection and eating of healthy diet for type 2 diabetes. Additionally, two-way text messages, will be sent to study participants to rate their ability on selection of food and eating of healthy diet based on the messages received after every 4 weeks. The combination of the one-way and two-way messages in this in the intervention arm are designed to increase engagement of the participants.

The control group will continue receiving standard care in the hospitals. This group shall also receive clinic appointment reminder text messages one day prior to the actual date.

Quantitative data will be analyzed by the intention to treat principle. Various patient characteristics and primary outcome measures, including anthropometric and biochemical measurements (HbA1c, Fasting Blood Glucose (FBG), lipid profiles) at baseline will be summarized using descriptive statistics. The descriptive statistics will include means and standard deviations for continuous variables and proportions for categorical variables.

HbA1c levels will be compared at 12 weeks between the two arms using an ANCOVA which will control for baseline HbA1c levels. The intervention and the control groups will be followed-up for six months to assess sustainability and mHealth satisfaction of the intervention. One-way and two-way text messaging data will be analyzed descriptively.

Subgroup analysis per hospital and participant socio-demographics including age, sex, education and income levels will be conducted. All statistical analyses will be performed using R version 4.0.3.

ELIGIBILITY:
Inclusion Criteria:

1. adults over the age of 18 years;
2. diagnosed the type 2 diabetes within the previous 1 year and obtaining care at a participating level 4 hospital;
3. able to read English or Swahili Language (self-reported).
4. currently own and able to read and send mobile text messages using any phone;

Exclusion Criteria:

1. are on dialysis;
2. are pregnant;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | 12 weeks
  Glycated hemoglobin in percentage (%)

SECONDARY OUTCOMES:
Fasting Plasma Glucose (FPG) | 12weeks
  Fasting Plasma Glucose in mg/dL
Total cholesterol (TC) | 12 Weeks
  Total blood cholesterol in mg/dL
Triglycerides (TG), | 12 Weeks
  Blood Triglycerides in mg/dL
High-density lipoprotein-cholesterol (HDL-C) | 12 Weeks
  High-density lipoprotein-cholesterol in mmol/L
mHealth (mobile health) Satisfaction | 12 Weeks
  User satisfaction shall use a 5-point likert scale from 1 (Strongly Disagree) to 5 (Strongly Agree. A score of 5 (Strongly Agree) means a high level of satisfaction, which is a better outcome. A low score of 1 (Strongly Disagree) means a low satisfaction level and therefore a worst outcome.
Weight | 12weeks
  Weight in meters
Height | 12 Weeks
  Height in Meters
Waist-hip ratio | 12 Weeks
  Waist-hip ratio in centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Jomo Kenyatta University of Agriculture and Technology, Nairobi, Kenya

DOCUMENTS (1):
  • Study Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT05013294/Prot_000.pdf